CLINICAL TRIAL: NCT06830837
Title: The Effect of Mandala Coloring on Anxiety and Depression Before Open Heart Surgery: a Randomized Controlled Trial
Brief Title: Mandala Coloring and Its Effect on Anxiety and Depression Before Open Heart Surgery
Acronym: Heart Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, MERVE KAYA, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AtaturkUnıverstynursing
Record Dates: First submitted 2025-02-12; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-12

CONDITIONS: Heart Surgery; Mandala Painting; Anxiety
Keywords: heart surgery; anxiety; mandala coloring; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention: Mandala coloring Grup 1 (Experimental): This group will color mandalas before the surgery.
  Interventions: Other: Mandala coloring
- No interventional: control grup Grup 2 (No Intervention): This group will not color mandalas before the surgery.

INTERVENTIONS:
Other: Mandala coloring — Eight pre-selected mandala drawings will be printed on separate A4 (21.0 cm × 29.7 cm) papers. After the patients are admitted to the hospital for the surgery process, the patients in the experimental group will be provided with at least 2 hours of mandala coloring per day until the day of their surgery. No intervention will be applied to the control group patients. Studies examining the effect of mandala coloring on reducing psychological symptoms have reported that using a circularly designed pattern in the mandala template, instead of a square design, has a greater effect on symptom management. Therefore, a circular-shaped mandala template will be used. Each participant will be provided with mandala coloring sheets and 12 colored pencils (red, orange, yellow, pink, light green, green, sky blue, blue, purple, brown, reddish-brown, and black) by the researcher.
  Other Names: mandala painting
  Arms: Intervention: Mandala coloring Grup 1

SUMMARY:
This study was conducted to determine the Effect of Mandala Coloring on Anxiety and Depression Before Open Heart Surgery. This was a randomized, controlled experimental study. The sample comprised 84 patients who underwent open heart surgery (control: 41; experimental: 43).

Eight pre-selected mandala drawings will be printed on separate A4 (21.0 cm × 29.7 cm) papers. After the patients are admitted to the hospital for the surgery process, the patients in the experimental group will be provided with at least 2 hours of mandala coloring per day until the day of their surgery. No intervention will be applied to the control group patients.

DETAILED DESCRIPTION:
Cardiovascular diseases are among the leading causes of death both globally and in our country. Despite advances in prevention, diagnosis, medical interventions, and surgical methods for heart diseases, "open heart surgery" remains one of the most effective methods in the treatment of cardiovascular disorders. For patients who do not respond to medical treatment, open heart surgery is often considered as a treatment option. Heart surgery is a surgical procedure that includes interventions on heart valves, repair of congenital defects, and coronary artery grafting. The surgical process is one of the most critical experiences in a patient's life, affecting them physically, psychologically, socially, and economically. Patients awaiting heart surgery experience high levels of anxiety and depression due to significant psychological stress, fear, worry, and uncertainties related to the surgery. For most patients, heart surgery is perceived as a crisis or a life-threatening event. When an individual faces a threatening event, it is cognitively assessed, and if deemed threatening, it triggers anxiety. Additionally, factors such as facing physically painful procedures, being away from family, losing a job, being in an unfamiliar environment, or encountering unknown devices can also contribute to anxiety during hospitalization.

Mandala is an art therapy technique that can provide psychological support and healing. This circular art has traditionally been used for meditation in various Asian cultures and symbolizes psychological wholeness. Mandala is a Sanskrit word meaning "circle, roundness, wholeness, and completion"; it provides mental calmness and relaxation. Mandala is used as a tool to enhance awareness, express oneself, solve negative problems, and promote healing. Mandala coloring is a safe and accessible activity that can be used as a complementary strategy to support mental health, requiring no special skills.

Through practices like mandala coloring, individuals project what they do not know onto the outside world and make it visible through this act of creation. The recovery process begins with this step. The artistic perspective of nursing involves understanding individuals' needs, identifying sources of anxiety and stress, and then developing practices that enhance people's abilities and competence, thus boosting their self-confidence and resilience. This study will be conducted to examine the effects of mandala coloring on anxiety and psychological well-being in patients undergoing open heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* Having no history of previous cardiothoracic surgery, eing newly diagnosed with CAD and registered on a wait list for CABG surgery, having literacy in the Turkish language

Exclusion Criteria:

* having a history of cognitive impairment, having other life-threatening medical conditions, such as cancer or stroke

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Surgical Anxiety Scale | 7 day before surgery
  The scale has three subdimensions: Health-Related Anxiety (items 7, 8, 9, 10, 12, and 13), Recovery-Related Anxiety (items 2, 14, 16, and 17), and Procedure-Related Anxiety (items 1, 3, 4, and 5). The total score of the Surgical Anxiety Scale (SAS) is obtained by summing the scores of the subdimension items and the three items not included in any subdimension. The lowest possible score on the scale is 0, and the highest score is 68. As the score increases, the level of surgical anxiety is considered higher.
Surgical Anxiety Scale | 1 day before surgery
  The scale has three subdimensions: Health-Related Anxiety (items 7, 8, 9, 10, 12, and 13), Recovery-Related Anxiety (items 2, 14, 16, and 17), and Procedure-Related Anxiety (items 1, 3, 4, and 5). The total score of the Surgical Anxiety Scale (SAS) is obtained by summing the scores of the subdimension items and the three items not included in any subdimension. The lowest possible score on the scale is 0, and the highest score is 68. As the score increases, the level of surgical anxiety is considered higher.
Surgical Anxiety Scale | On the day of surgery
  The scale has three subdimensions: Health-Related Anxiety (items 7, 8, 9, 10, 12, and 13), Recovery-Related Anxiety (items 2, 14, 16, and 17), and Procedure-Related Anxiety (items 1, 3, 4, and 5). The total score of the Surgical Anxiety Scale (SAS) is obtained by summing the scores of the subdimension items and the three items not included in any subdimension. The lowest possible score on the scale is 0, and the highest score is 68. As the score increases, the level of surgical anxiety is considered higher.
Hospital Anxiety and Depression Scale | 7 day before surgery
  The scale consists of 14 items, and it has two subdimensions: anxiety and depression. Seven items (odd numbers) measure anxiety, and seven items (even numbers) measure depression. The scale uses a 4-point Likert format, with scores ranging from 0 to 3. Each item on the scale has a different scoring method. Items 1, 3, 5, 6, 8, 10, 11, and 13 are reverse-scored, while items 2, 4, 7, 9, 12, and 14 are scored normally.
  For the anxiety subdimension, the items 1, 3, 5, 7, 9, 11, and 13 are used; for the depression subdimension, the items 2, 4, 6, 8, 10, 12, and 14 are used. Patients can score between 0 and 21 on each subdimension. The cutoff point for anxiety is 10, and the cutoff point for depression is 7. Patients who score above these cutoff points are considered at risk.
Hospital Anxiety and Depression Scale | 1 day before surgery
  The scale consists of 14 items, and it has two subdimensions: anxiety and depression. Seven items (odd numbers) measure anxiety, and seven items (even numbers) measure depression. The scale uses a 4-point Likert format, with scores ranging from 0 to 3. Each item on the scale has a different scoring method. Items 1, 3, 5, 6, 8, 10, 11, and 13 are reverse-scored, while items 2, 4, 7, 9, 12, and 14 are scored normally.
  For the anxiety subdimension, the items 1, 3, 5, 7, 9, 11, and 13 are used; for the depression subdimension, the items 2, 4, 6, 8, 10, 12, and 14 are used. Patients can score between 0 and 21 on each subdimension. The cutoff point for anxiety is 10, and the cutoff point for depression is 7. Patients who score above these cutoff points are considered at risk.
Hospital Anxiety and Depression Scale | On the day of surgery
  The scale consists of 14 items, and it has two subdimensions: anxiety and depression. Seven items (odd numbers) measure anxiety, and seven items (even numbers) measure depression. The scale uses a 4-point Likert format, with scores ranging from 0 to 3. Each item on the scale has a different scoring method. Items 1, 3, 5, 6, 8, 10, 11, and 13 are reverse-scored, while items 2, 4, 7, 9, 12, and 14 are scored normally.
  For the anxiety subdimension, the items 1, 3, 5, 7, 9, 11, and 13 are used; for the depression subdimension, the items 2, 4, 6, 8, 10, 12, and 14 are used. Patients can score between 0 and 21 on each subdimension. The cutoff point for anxiety is 10, and the cutoff point for depression is 7. Patients who score above these cutoff points are considered at risk.

IPD SHARING:
Plan to Share IPD: No